CLINICAL TRIAL: NCT05816928
Title: Ventilation-Perfusion Matching in Early-stage Prone Position Ventilation: A Comparison Between COVID-19 ARDS and ARDS From Other Etiologies
Brief Title: Ventilation-Perfusion Matching in Early-stage Prone Position Ventilation
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EIT20230403
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; ICU; COVID19; Electrical impedance tomography
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID19-associated ARDS (CARDS): This group included COVID19 patients with acute respiratory distress syndrome. Patients were put under prone position while their pulmonary function was measured using EIT before and after proning.
- Non-COVID19-associated ARDS (non-CARDS): This group included patients with acute respiratory distress syndrome from other etiologies. Patients were put under prone position while their pulmonary function was measured using EIT before and after proning.

SUMMARY:
Prone positioning has been widely used in critical care medicine to improve oxygenation in patients with acute respiratory distress syndrome (ARDS). This study aimed to compare the effect of pronation on lung ventilation-perfusion matching between COVID19-associated acute respiratory distress syndrome (CARDS) and ARDS from other etiologies (non-CARDS) using electrical impedance tomography (EIT).

DETAILED DESCRIPTION:
In this prospective study, both COVID19-associated ARDS (CARDS) patients and patients with ARDS from other etiologies (non-CARDS) were enrolled. Electrical impedance tomography (EIT) was used to evaluate the changes in ventilation and perfusion between supine and prone positions. Baseline values of the area of DeadSpace, shunt, ventilation-perfusion matching (VQmatch) were identified at the time of enrollment. Within the defined VQmatch region, the global inhomogeneity index (VQmatch-GI) was calculated to assess the degree of uniformity within the region. Prone position was applied immediately after the baseline data were collected. After 2 hours of proning, another EIT examination was conducted. Parameters such as DeadSpace, shunt, VQmatch, and other common measurements before and after pronation were taken and compared to evaluate the effect of prone positioning on CARDS and non-CARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* Diagnosed with ARDS based on the Berlin Definition of ARDS
* Under mechanical ventilation

Exclusion Criteria:

* Contraindications to EIT examination and prone position
* Refusal of signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes COVID19-associated ARDS patients and ARDS patients of other etiologies in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
DeadSpace | 3 months
  The area of Deadspace will be assessed using electrical impedance tomography
Shunt | 3 months
  Shunt will be assessed using electrical impedance tomography
Ventilation-perfusion matching (VQmatch) | 3 months
  VQmatch will be assessed using electrical impedance tomography
Global inhomogeneity index (VQmatch-GI) | 3 months
  Within the defined VQmatch region assessed by electrical impedance tomography, the global inhomogeneity index (VQmatch-GI) was calculated to assess the degree of uniformity within the region.

SECONDARY OUTCOMES:
Ventilation | 3 months
  The ventilation of the lungs is assessed by electrical impedance tomography before and after prone positioning.
Perfusion | 3 months
  The perfusion of the lungs is assessed by electrical impedance tomography before and after prone positioning.
Center of Ventilation (CoV) | 3 months
  The center of ventilation of the lungs is assessed by electrical impedance tomography before and after prone positioning.
Standard deviation of regional ventilation delay | 3 months
  The standard deviation of regional ventilation delay of the lungs is assessed by electrical impedance tomography before and after prone positioning.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, MD, Principal Investigator — Peking Union Medical College
Locations (1):
- PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Li H, Chi Y, Frerichs I, Zhao Z, Li Y, Zhang C, Chu H, He H, Long Y. Ventilation-perfusion matching in early-stage of prone position ventilation: a prospective cohort study between COVID-19 ARDS and ARDS from other etiologies. Physiol Meas. 2025 Jan 29;13(1). doi: 10.1088/1361-6579/ada8f1. PMID 39793207